CLINICAL TRIAL: NCT05538416
Title: Short-term Clinical Outcome of Cortical Bone Trajectory Compared With the Traditional "Open" and Minimal Invasive Posterior Lumbar Interbody Fusion
Status: Recruiting | Type: Observational
Sponsor: Jos M. A. Kuijlen (Other)
Responsible Party: Sponsor-Investigator, Jos M. A. Kuijlen, Dr. MD, PhD, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Other Study IDs: UMCG202200129
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Degenerative Spondylolisthesis; Spondylolytic Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open PLIF: Patients undergoing conventional open posterior lumbar interbody fusion (PLIF) surgery. A long midline skin incision (10-15 cm) is made, after which the paravertebral muscles are detached from the midline and retracted laterally in order to expose the facet joints and pedicle entry point. After the pedicle screws are positioned, the disc will be removed bilaterally and packed with autogenous bone chips, followed by bilateral placement of polyetheretherketone (PEEK) PLIF cages.
  Interventions: Procedure: Posterior Lumbar Interbody Fusion (PLIF)
- CBT-PLIF: Patient undergoing minimal access PLIF surgery with cortical bone trajectory (CBT-PLIF). The CBT-PLIF uses more medialized entry points, closer to the spinal process. Due to the medial approach of this technique, a smaller incision is needed and the need to retract muscles laterally is minimalized.
  Interventions: Procedure: Posterior Lumbar Interbody Fusion (PLIF)
- MI-PLIF: Patients undergoing minimal invasive PLIF surgery. A small midline incision (3-5 cm) will be made to perform mini-open decompression and placement of bilateral PEEK PLIF cages. In addition, two small paramedian incisions will be made on both sides for percutaneous pedicle screw fixation.
  Interventions: Procedure: Posterior Lumbar Interbody Fusion (PLIF)

INTERVENTIONS:
Procedure: Posterior Lumbar Interbody Fusion (PLIF) — Spinal fusion in the lumbar spine by inserting a cage directly into the disc space. This is an observational study in which the standard procedure/care is followed.

SUMMARY:
A combined prospective cohort study and retrospective analysis of previously collected data. Three different techniques for posterior lumbar interbody fusion (PLIF) are compared: CBT-PLIF, MI-PLIF and open PLIF. A total of 180 patients are included, who will be followed up to 6 weeks postoperatively.

DETAILED DESCRIPTION:
A combined prospective cohort study for CBT-PLIF and retrospective analysis of prospectively collected data from the MISOS study, regarding traditional open PLIF and MI-PLIF. A total of 180 patients will be included in the study: 60 prospective CBT-PLIF patients, 60 retrospective open PLIF patients and 60 retrospective MI-PLIF patients.

The new data will be collected prospectively by means of questionnaires. No biomaterial will be collected. The included patients will be asked to complete questionnaires before surgery, 2 and 6 weeks after surgery. In addition, VAS scores will be noted throughout the hospital stay, 2 and 6 weeks after surgery.

Inclusion criteria: Patients aged 18-75 years with neurogenic claudication and/or radicular leg pain due to low-grade (Meyerding grades l and ll) degenerative or spondylolytic spondylolisthesis with persistent symptoms for more than 3 months.

Exclusion criteria: previous spinal fusion surgery at the same level, osteoporosis (only when using bisphosphonate), active infection or previous infection at the surgical site, active cancer, spondylolisthesis grade III or greater, more than one symptomatic level requiring fusion, pregnancy, contraindication to surgery, severe mental or psychiatric disorder, substance abuse, insufficient knowledge of the Dutch language and morbid obesity (body mass index >40).

Main research question: Does the CBT-PLIF provide less low back pain in the short term than the traditional open PLIF and the MI-PLIF?

Primary outcome measure

* Low back pain measured with the Visual Analogue Scale (VAS) 2 weeks after surgery Secondary Outcomes
* Low back pain during hospitalization (measured every day), 2 and 6 weeks after surgery
* Leg pain
* Oswestry Disability Index
* Quality of life (EQ-5D-5L)
* Observed patient recovery
* Other parameters such as complications, surgical parameters (intraoperative blood loss, duration of surgery), length of stay in hospital and return to work

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* Degenerative or spondylolytic spondylolisthesis
* Neurogenic claudication and/or radicular leg pain
* Low grade (Meyerding grade l and ll)
* Persistent complaints for over 3 months

Exclusion Criteria:

* Previous spine fusion surgery at the same level
* Osteoporosis
* Active infection or prior infection at the surgical site
* Active cancer
* Spondylolisthesis grade lll or greater
* More than one symptomatic level that needs fusion
* Pregnancy
* Contraindication for surgery
* Severe mental or psychiatric disorder
* Substance abuse
* Inadequate knowledge of Dutch language
* Morbid obesity (body mass index >40)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 180 participants, 60 prospective CBT-PLIF participants, 60 retrospective open-PLIF and 60 retrospective MI-PLIF participants. Patients aged 18-75 years with neurogenic claudication and/or radicular leg pain due to a low grade (Meyerding grade l and ll) degenerative or spondylolytic spondylolisthesis with persistent complaints for over 3 months will be included in the study. Patients are operated in either the University Medical Centre Groningen (UMCG) or in the Haaglanden Medical Centre (HMC).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
VAS low back pain | 2 weeks postoperative
  VAS for low back pain ranging from 0mm (no pain) to 100mm (worst pain imaginable)

SECONDARY OUTCOMES:
VAS low back pain | During hospital stay, measured each day and 6 weeks postoperative
  VAS for low back pain ranging from 0mm (no pain) to 100mm (worst pain imaginable)
VAS leg pain | During hospital stay, measured each day, 2 and 6 weeks postoperative
  VAS for leg pain ranging from 0mm (no pain) to 100mm (worst pain imaginable)
Oswestry Disability Index | 2 and 6 weeks postoperative
  Used to quantify the degree of functional impairment in patients with low back pain. Ranging from 0 (no disability) to 100 (bed bound)
Quality of Life (QoL) | 2 and 6 weeks postoperative
  Measured by the EQ-5D-5L
Perceived recovery of the patient | 2 and 6 weeks postoperative
  scored on a 7-Likert scale, with scores ranging from 'worse than ever' to 'complete recovery'

CONTACTS AND LOCATIONS:
Overall Officials: Jos M.A. Kuijlen, MD, PhD, Principal Investigator — University Medical Centre Groningen (UMCG), Hanzeplein 1, 9713GZ Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No